CLINICAL TRIAL: NCT06586229
Title: Screening and Management of Hyperuricemia in Patients with Chronic Medical Diseases in Assiut University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Huda Abdelkader, principal investigator, Assiut University
Other Study IDs: screening of hyperuricmia
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this study, we aimed to evaluate patients with chronic medical diseases in Assiut university hospitals for -Detection of asymptomatic hyperuricemia .

* Early identification of associated comorbidities .
* Management of indicated hyperurecimia .

DETAILED DESCRIPTION:
Hyperuricemia is classically defined as a serum uric acid (SUA) of more than 7.0 mg/dL in men or more than 6.0 mg/dL in women . Asymptomatic hyperuricemia is a condition, where patients have elevated levels of SUA, yet do not exhibit symptoms or signs of monosodium urate crystal deposition, such as gout attacks, urolithiasis, or uric acid nephropathy . SUA can be elevated 10 to 15 years before clinical manifestations of gout . Up to 21% of the general population and 25% of hospitalized patients are estimated to have asymptomatic hyperuricemia .

Uric acid excretion mostly occurs via the kidneys, so decreased glomerular filtration rates in chronic kidney (CKD) patients contribute to the population increase in hyperuricemia. Conversely, studies suggest that hyperuricemia may contribute to CKD , raising the possibility that urate-lowering therapies (ULTs) could be useful in slowing CKD progression . There was no independent association between hyperuricemia and systemic arterial hypertension. Also, hyperuricemia has been reported as an independent risk factor for both coronary artery disease, congestive heart failure and diabetes mellitus.

So efforts should be made to recognize individuals at risk of hyperuricemia by evaluating dietary habits, family history, and lifestyle factors, and regularly monitor SUA levels. As well as, management strategies, including lifestyle modifications, pharmacotherapy, and dietary interventions, to effectively control SUA and reduce the risk of associated complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older who were diagnosed with chronic medical diseases as diabetes mellitus , hypertension , obesity , metabolic syndrome , chronic kidney disease and cardiovascular disease (ischemic cardiomyopathy, heart failure ,coronary arteries disease) .

Exclusion Criteria:

* patients under the age of 18.
* patients kown to have gouty arthritis
* patients with acute kidney disease .
* patients receiving thiazide diuretics.
* patients with tumour lysis syndrome .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The estimated minimum required sample size is 61 patients in one group
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
screening for asymptomatic hyperuricaemia | baseline
  Detection of asymptomatic hyperuricemia patients with chronic medical diseases. Early identification of associated comorbidities . Management of indicated hyperurecimia .

CONTACTS AND LOCATIONS:
Overall Officials: Huda Abdelkader Khalafallah, Principal Investigator — Assiut University; Mohammed Abbas Sobh, Study Director — Assiut University; Ayat Salah Ahmed, Study Director — Assiut University